CLINICAL TRIAL: NCT02828033
Title: A Pilot Trial of Rilonacept for Treatment of Autoimmune Neurosensory Hearing Loss
Brief Title: Rilonacept for Treatment of Autoimmune Neurosensory Hearing Loss
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanley Cohen (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Stanley Cohen, MD, Metroplex Clinical Research
Organization: Metroplex Clinical Research (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rilonacept IIS 1604
Record Dates: First submitted 2016-07-01; First posted 2016-07-11 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Autoimmune Neurosensory Hearing Loss (ANSHL)
MeSH Terms: interventions — rilonacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rilonacept (Experimental): A loading dose of 320 mg the first dose then be a once-weekly injection of 160 mg for 24 weeks
  Interventions: Drug: Rilonacept

INTERVENTIONS:
Drug: Rilonacept — All patients will receive rilonacept with an initial loading dose of 320 mg delivered as two, 2-mL, subcutaneous injections of 160 mg each given on the same day at two different sites. The initial dose will be administered at the study site by study personnel. Dosing will then be a once-weekly injection of 160 mg administered as a single, 2-mL, subcutaneous injection by the patient at home. Patients will be dosed for 24 weeks.
  Other Names: IL-1 Trap; Arcalyst

SUMMARY:
This study is an open label proof of concept study of rilonacept for patients with ANSHL

DETAILED DESCRIPTION:
Ten (10) patients in total will be enrolled in this study at Metroplex Clinical Research Center in Dallas, TX. Patients may be identified and referred by local area audiologist. The ANSHL study population will be defined by inclusion and exclusion criteria designed to limit enrollment to individuals with idiopathic, progressive, bilateral sensorineural hearing loss, to ensure appropriate candidates for treatment with study medications, and to identify those with a high likelihood of complying with the study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of progressive sensironeural hearing loss greater than or equal to 30 dB in both ears at one or more frequencies (250, 500, 1000, 2000, 3000, 4000, 6000 or 8000 Hz) and idiopathic-based on clinical evaluation, blood tests, and radiographic imaging.
2. Documented improvement in hearing by audiogram after 30 days of treatment with high dose prednisone 40-60 mg/d. Improvement is defined by 10 dB improvement in pure tone average (500-3000 dB) or an improvement in word identification score of at least 12% in either ear (both relative to baseline). Prednisone could be started at screening but patients may have received prednisone prior to screening and the pre prednisone audiogram will be used as the screening audiogram for this study. It is expected the majority of these patients will screen for the study in this fashion as they are referred from otoloaryngology after initial treatment.
3. 18-75 years of age
4. Able and willing to give written informed consent and comply with the requirements of the study protocol
5. Negative serum pregnancy test (for women of child bearing potential). Males and Females of child bearing potential must agree to consistently use 2 forms of highly effective birth control (at least 1 of which must be a barrier method) starting at screening and throughout the study period and for 3 months after the final study drug administration.

Exclusion Criteria:

1. Pregnant or nursing, or planning to become pregnant or father a child within 3 months after receiving the last dose of study drug
2. Have a known or suspected current active infection or a history of chronic or recurrent infectious disease including, but not limited to, chronic renal infection, chronic chest infections, chronic sinusitis, recurrent urinary tract infections, an open, draining, infected skin wound.
3. Within 2 months of first study drug administration, have had a serious infection, have been hospitalized for an infection, have been treated with PO antibiotics for longer than 2 weeks, or have been treated with intravenous (IV) antibiotics for an infection
4. Uncontrolled diabetes at the baseline visit (defined as HbA1c ≥9.0%)
5. Patients requiring dialysis
6. Patients who have had an organ transplant
7. Treatment with any systemic {non-glucocorticoid} immunosuppressants (e.g. methotrexate, azathioprine, cyclosporine, mercaptopurine, mycophenolate mofetil, tacrolimus, sirolimus within 4 weeks of baseline rilonacept administration. No leflunomide treatment within 8 weeks prior to baseline administration. No etanercept, adalimumab, infliximab, tocilizumab, abatacept, or natalizumab, within 2 months prior to baseline visit; No rituxan for 12 months prior to baseline and evidence of normal B cell count required. Patients previously treated with anakinra for ANSHL cannot be enrolled.
8. Prohibited Medications:

   1. Strong CYP3A4 inhibitors, protease inhibitors or P-gp inhibitors.
   2. Long-acting or extended release forms of opiates.
   3. Live or live-attenuated vaccines are excluded during the course of the study
   4. IA and IM glucocorticoid injections. Long-acting steroid preparations are not allowed during study (this includes suspensions and all forms of dexamethasone).
9. History of a demyelinating disease or symptoms suggestive of multiple sclerosis
10. Treatment with a live or live-attenuated virus vaccine during the 3 months prior to baseline
11. Estimated glomerular filtration rate (eGFR) of <20 mL/min/1.73m2 or patients planning to start dialysis within a year from the screening visit
12. Baseline laboratory test results meeting any of the following criteria:

    1. Hemoglobin (Hgb)<8.5 g/dL (85 g/L)
    2. Neutrophil count<1.5 x 103/μL
    3. Platelet count<100 x 103/μL
    4. Total bilirubin exceeding 1.5 times the upper limit of normal (ULN) unless consistent with Gilbert's syndrome
    5. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) exceeding 2 times the ULN
13. Positive history of human immunodeficiency virus (HIV) by clinical or serological testing.
14. Presence of hepatitis B surface antigen (HBsAg) and/or hepatitis C antibody (HCV) by serologic testing
15. History of active TB prior to screening or chest x-ray showing evidence of malignancy or any abnormalities suggestive of prior tuberculosis (TB) infection, including, but not limited to, apical scarring, apical fibrosis, or multiple calcified granulomata.
16. A positive intradermal skin tuberculin test (purified protein derivative [PPD] 5 tuberculin unit [TU]) of ≥5 mm induration read at 48 to 72 hours or positive QuantiFERON-gold testing. Signs or symptoms suggestive of active TB (e.g. new cough lasting >14 days or a change in chronic cough, persistent fever, unintentional weight loss, night sweats) upon review of medical history and/or physical examination. If the patient is thought to have a false-positive PPD because of prior BCG vaccination and it is known that the patient has been negative on testing obtained outside the protocol for M. tuberculosis infection using a cell-based interferon gamma assay the patient is eligible for enrollment.
17. Recent close contact with a person with active TB
18. History of latent untreated TB. Patients who have been adequately treated for latent TB are eligible for enrollment.
19. Any other medical condition that in the opinion of the investigator could adversely affect the patient's participation or interfere with evaluations. This includes significant concomitant illness such as, but not limited to, cardiac, renal, neurological, endocrinological, metabolic, pulmonary, gastrointestinal, or psychiatric disease.
20. History or presence of malignancy within 5 years of the screening visit (other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix)
21. History of a myeloproliferative disorder
22. History of alcohol abuse within last 5 years or current intake of 21 or more alcohol-containing drinks per week
23. History of drug abuse within the 5 years prior to screening
24. Patients with previous exposure to rilonacept
25. Use of any investigational drug within 30 days or within 5 half-lives (whichever is longer) prior to the screening visit
26. Sexually active men or women of childbearing potential who are unwilling to practice adequate contraception during the study (adequate contraceptive measures are defined as the use of two highly effective forms of birth control, include stable use of oral contraceptives or other prescription pharmaceutical contraceptives; intrauterine device; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly)
27. Known moderate-to-severe liver disease (Child-Pugh class B or C)
28. Known hypersensitivity to CHO cell derived therapeutics or proteins or any components of rilonacept

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Improvement in hearing in comparison to baseline values | 24 weeks
  1. An improvement in pure tone average (500 to 3000 Hz) by 10 dB in at least one ear or
  2. An improvement of word identification score of at least 12 percent; both relative to baseline values

SECONDARY OUTCOMES:
Pt reported evaluation of auditory acuity | 24 weeks
  Pt reported evaluation of auditory acuity as measured on a 0-100 Visual Analog Scale (VAS). Patients with a 25% improvement in VAS will be considered responders.
Vertigo evaluation | 24 weeks
  Vertigo will be evaluated using the validated OTA Dizziness Handicap Inventory (DHI). A change in category is considered clinically significant.
Tinnitus evaluation | 24 weeks
  Tinnitus will be evaluated using the validated OTA Tinnitus Handicap Inventory (THI). A change of 6 points on this scale is considered clinically meaningful.
Quality of Life assessment | 24 weeks
  Validated auditory quality of life questionnaire- Response is defined as a 5% or greater improvement

CONTACTS AND LOCATIONS:
Overall Officials: Stanley B Cohen, MD, Principal Investigator — Metroplex Clinical Research Center
Locations (1):
- Metroplex Clinical Research Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Outcomes data

REFERENCES:
- [Background] McCabe BF. Autoimmune sensorineural hearing loss. Ann Otol Rhinol Laryngol. 1979 Sep-Oct;88(5 Pt 1):585-9. doi: 10.1177/000348947908800501. PMID 496191
- [Background] Harris JP, Sharp PA. Inner ear autoantibodies in patients with rapidly progressive sensorineural hearing loss. Laryngoscope. 1990 May;100(5):516-24. doi: 10.1288/00005537-199005000-00015. PMID 2329911
- [Background] Moscicki RA, San Martin JE, Quintero CH, Rauch SD, Nadol JB Jr, Bloch KJ. Serum antibody to inner ear proteins in patients with progressive hearing loss. Correlation with disease activity and response to corticosteroid treatment. JAMA. 1994 Aug 24-31;272(8):611-6. PMID 8057517
- [Background] Tebo AE, Szankasi P, Hillman TA, Litwin CM, Hill HR. Antibody reactivity to heat shock protein 70 and inner ear-specific proteins in patients with idiopathic sensorineural hearing loss. Clin Exp Immunol. 2006 Dec;146(3):427-32. doi: 10.1111/j.1365-2249.2006.03227.x. PMID 17100761
- [Background] Hirose K, Wener MH, Duckert LG. Utility of laboratory testing in autoimmune inner ear disease. Laryngoscope. 1999 Nov;109(11):1749-54. doi: 10.1097/00005537-199911000-00005. PMID 10569401
- [Background] Bouman H, Klis SF, Meeuwsen F, de Groot JC, Smoorenburg GF, Veldman JE. Experimental autoimmune inner ear disease: an electrocochleographic and histophysiologic study. Ann Otol Rhinol Laryngol. 2000 May;109(5):457-66. doi: 10.1177/000348940010900504. PMID 10823474
- [Background] McCabe BF. Autoimmune inner ear disease: therapy. Am J Otol. 1989 May;10(3):196-7. PMID 2750868
- [Background] Saracaydin A, Katircioglu S, Katircioglu S, Karatay MC. Azathioprine in combination with steroids in the treatment of autoimmune inner-ear disease. J Int Med Res. 1993 Jul-Aug;21(4):192-6. doi: 10.1177/030006059302100404. PMID 8112477
- [Background] Sismanis A, Wise CM, Johnson GD. Methotrexate management of immune-mediated cochleovestibular disorders. Otolaryngol Head Neck Surg. 1997 Feb;116(2):146-52. doi: 10.1016/S0194-59989770316-4. PMID 9051055
- [Background] Luetje CM. Theoretical and practical implications for plasmapheresis in autoimmune inner ear disease. Laryngoscope. 1989 Nov;99(11):1137-46. doi: 10.1288/00005537-198911000-00006. PMID 2811552
- [Background] Kitashara M, Yazawa.Y, Uchida K. Immunoglobulin treatment for advance cases of bilateral Meniere's disease. In: Nadol JB ed. Meniere's disease: pathogenesis, pathophysiology, diagnosis and treatment. Berkeley, Ca: Kugler Publications; 1989; 411-419.
- [Background] Harris JP, Weisman MH, Derebery JM, Espeland MA, Gantz BJ, Gulya AJ, Hammerschlag PE, Hannley M, Hughes GB, Moscicki R, Nelson RA, Niparko JK, Rauch SD, Telian SA, Brookhouser PE. Treatment of corticosteroid-responsive autoimmune inner ear disease with methotrexate: a randomized controlled trial. JAMA. 2003 Oct 8;290(14):1875-83. doi: 10.1001/jama.290.14.1875. PMID 14532316
- [Background] Broughton SS, Meyerhoff WE, Cohen SB. Immune-mediated inner ear disease: 10-year experience. Semin Arthritis Rheum. 2004 Oct;34(2):544-8. doi: 10.1016/j.semarthrit.2004.07.001. PMID 15505770
- [Background] Cohen S, Shoup A, Weisman MH, Harris J. Etanercept treatment for autoimmune inner ear disease: results of a pilot placebo-controlled study. Otol Neurotol. 2005 Sep;26(5):903-7. doi: 10.1097/01.mao.0000185082.28598.87. PMID 16151336
- [Background] Rahman MU, Poe DS, Choi HK. Etanercept therapy for immune-mediated cochleovestibular disorders: preliminary results in a pilot study. Otol Neurotol. 2001 Sep;22(5):619-24. doi: 10.1097/00129492-200109000-00010. PMID 11568668
- [Background] Cohen S, Roland P, Shoup A, Lowenstein M, Silverstein H, Kavanaugh A, Harris J. A pilot study of rituximab in immune-mediated inner ear disease. Audiol Neurootol. 2011;16(4):214-21. doi: 10.1159/000320606. Epub 2010 Oct 27. PMID 20980741
- [Background] Rynne M, Maclean C, Bybee A, McDermott MF, Emery P. Hearing improvement in a patient with variant Muckle-Wells syndrome in response to interleukin 1 receptor antagonism. Ann Rheum Dis. 2006 Apr;65(4):533-4. doi: 10.1136/ard.2005.038091. PMID 16531551
- [Background] Yamazaki T, Masumoto J, Agematsu K, Sawai N, Kobayashi S, Shigemura T, Yasui K, Koike K. Anakinra improves sensory deafness in a Japanese patient with Muckle-Wells syndrome, possibly by inhibiting the cryopyrin inflammasome. Arthritis Rheum. 2008 Mar;58(3):864-8. doi: 10.1002/art.23261. PMID 18311804
- [Background] Pathak S, Goldofsky E, Vivas EX, Bonagura VR, Vambutas A. IL-1beta is overexpressed and aberrantly regulated in corticosteroid nonresponders with autoimmune inner ear disease. J Immunol. 2011 Feb 1;186(3):1870-9. doi: 10.4049/jimmunol.1002275. Epub 2011 Jan 3. PMID 21199898
- [Background] Vambutas A, Lesser M, Mullooly V, Pathak S, Zahtz G, Rosen L, Goldofsky E. Early efficacy trial of anakinra in corticosteroid-resistant autoimmune inner ear disease. J Clin Invest. 2014 Sep;124(9):4115-22. doi: 10.1172/JCI76503. Epub 2014 Aug 18. PMID 25133431